CLINICAL TRIAL: NCT02204644
Title: Randomized, Multi-center, Open-label Phase III Study of the Efficacy and Safety of Flumatinib vs Imatinib as First Line Treatment in Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia.
Brief Title: The Study of the Efficacy and the Safety of Flumatinib vs Imatinib as First Line Treatment in Patients With CML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10096-301
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2014-07

CONDITIONS: CML, CML-CP,MMR,TKI
MeSH Terms: interventions — flumatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flumatinib mesylate tablets (Experimental): Flumatinib mesylate tablets 600mg qd for 12 months
  Interventions: Drug: Flumatinib 600mg qd
- Imatinib mesylate tablets (Active Comparator): Imatinib mesylate tablets 400mg qd for 12months
  Interventions: Drug: Imatinib 400mg qd

INTERVENTIONS:
Drug: Flumatinib 600mg qd
  Arms: Flumatinib mesylate tablets
Drug: Imatinib 400mg qd
  Arms: Imatinib mesylate tablets

SUMMARY:
A study to observe the efficacy and the safety of Flumatinib vs Imatinib as first line treatment in patients with newly diagnosed chronic phase chronic myelogenous leukemia.

Randomized,Open Label,Control

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75 year-old
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
3. Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase (Ph + CP-CML) within 6 months of diagnosis
4. Adequate organ function

Exclusion Criteria:

1. received TKIs drug treatment before enrollment
2. Central nervous system leukemia
3. Previous anti-CML therapy over two weeks (hydroxyurea, except anagrelide) or surgery (including hematopoietic stem cell transplantation)
4. Cardiac dysfunction
5. Previous splenectomy
6. History of congenital or acquired bleeding disorders unrelated to CML
7. Previous malignancy except CML
8. Acute or chronic liver or severe kidney disease unrelated to CML
9. Pregnant, breastfeeding, child bearing potential but failed to take effective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
SIX-month major molecular response rate | six months

SECONDARY OUTCOMES:
major molecular response rate | 3 months, 9 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Blood Diseases, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhang L, Meng L, Liu B, Zhang Y, Zhu H, Cui J, Sun A, Hu Y, Jin J, Jiang H, Zhang X, Li Y, Liu L, Zhang W, Liu X, Gu J, Qiao J, Ouyang G, Liu X, Luo J, Jiang M, Xie X, Li J, Zhao C, Zhang M, Yang T, Wang J. Flumatinib versus Imatinib for Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia: A Phase III, Randomized, Open-label, Multi-center FESTnd Study. Clin Cancer Res. 2021 Jan 1;27(1):70-77. doi: 10.1158/1078-0432.CCR-20-1600. Epub 2020 Sep 14. PMID 32928796